CLINICAL TRIAL: NCT02949024
Title: Open-Label Study of the Safety and Efficacy of Suprachoroidal CLS-TA Alone or in Combination With Intravitreal Aflibercept for the Treatment of Diabetic Macular Edema
Brief Title: Suprachoroidal Injection of CLS-TA Alone or With Aflibercept in Subjects With Diabetic Macular Edema
Acronym: HULK
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clearside Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLS1004-101; NCT02944240 (obsolete NCT alias)
Record Dates: First submitted 2016-10-25; First posted 2016-10-31 (Estimated); Results first posted 2021-04-19 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetes mellitus; Diabetic retinopathy; Microneedle; Microinjection; Triamcinolone; Choroid; Choroid Injection; Aflibercept; Suprachoroidal; Triamcinolone acetonide
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy | interventions — aflibercept; Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TX Naïve Arm (Experimental): Treatment in the TX Naive arm will consist of one unilateral injection of IVT aflibercept in combination with one unilateral injection of SC CLS-TA in the same eye.
  Interventions: Drug: IVT Aflibercept; Drug: SC CLS-TA
- Previous TX Arm (Experimental): Treatment in the Previous TX arm of the study will consist of one unilateral injection of SC CLS-TA.
  Interventions: Drug: SC CLS-TA

INTERVENTIONS:
Drug: IVT Aflibercept — IVT aflibercept [2 mg (50 µL)]
  Other Names: Aflibercept
  Arms: TX Naïve Arm
Drug: SC CLS-TA — [4 mg (100 µL)]
  Other Names: Triamcinolone Acetonide

SUMMARY:
This study is designed to demonstrate the safety and tolerability of suprachoroidal CLS-TA alone or in combination with intravitreal aflibercept in subjects with diabetic macular edema associated with diabetes mellitus.

DETAILED DESCRIPTION:
This is a Phase 1/2, multicenter, open-label study in subject with DME associated with diabetes mellitus.

Subjects will be screened and if eligible, will be assigned to study arm at the Baseline Visit (Visit 1, Day 0).

Following the Baseline Visit, subjects will participate in six monthly follow-up visits (Visit 2-7; Weeks 4-24) for safety and efficacy assessments and to determine whether additional therapy is needed based upon pre-defined criteria.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 years of age with type 1 or type 2 diabetes mellitus
* DME with central involvement (>320 microns in the central subfield on SD-OCT) in the study eye
* ETDRS BCVA letter score of 83 to 14, inclusive (Snellen equivalent of 20/25 to 20/500) in the study eye

Exclusion Criteria:

* Evidence of DME due to any other cause other than diabetes mellitus in the study eye
* PRP or focal laser photocoagulation in the study eye within 90 days of screening
* Intraocular pressure ≥ 22 mmHg or uncontrolled glaucoma (open angle or angle closure) in the study eye
* History of any previous ophthalmic surgeries in the study eye within 90 days of screening
* High risk PDR in the study eye, for whom enrollment into the study, in the principal investigator's opinion would put the eye at undue risk for vision loss
* Any previous treatment in the study eye with ILUVIEN implant
* Previous treatment for DME in the study eye (TX naive arm only); treatment in the study eye for DME greater than 1 year prior to screening can be considered as treatment naive, at the investigator's discretion
* Subjects previously treated for DME cannot have been treated in the study eye with an intravitreal injection of anti-VEGF or periocular corticosteroids within 90 days prior to screening (Previous TX arm only)
* Subjects previously treated for DME cannot have been treated in the study eye with intraocular corticosteroids within 6 months prior to screening (Previous TX arm only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ciulla, MD MBA, Study Director — Clearside Biomedical, Inc.
Locations (2):
- United States (2):
  - Retina Vitreous Associates Medical Group Inc, Mountain View, California
  - Retina Consultants of Houston, PA, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TX Naïve Arm | Previous TX Arm
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat population included all subjects who received study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | TX Naïve Arm | Previous TX Arm | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age of patients in years relative to the date of the Screening visit.
  Years | 61.9 (7.28) | 63.1 (8.31) | 62.5 (7.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Baseline Best Corrected Visual Acuity [Mean (Standard Deviation); unit: Letters] — Best corrected visual acuity (BCVA) refers to the measurement of the best possible vision that can be achieved following refraction or correction. BCVA was assessed following the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol and was measured as the number of letters read correctly on an ETDRS eye chart.
  Letters | 67.2 (11.66) | 67.2 (8.95) | 67.2 (10.12)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events and Serious Adverse Events
Description: Number of participants with treatment emergent adverse events and serious adverse events reported over 6 months of follow-up
Time Frame: Over 6 months of follow-up
Population: The Safety population included all subjects who received study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | TX Naïve Arm | Previous TX Arm
Number analyzed (Participants) | 10 | 10
Participants
  Number of participants with treatment emergent adverse events | 8 | 9
  Number of participants with serious adverse events | 0 | 0

2. Secondary Outcome: Mean Change From Baseline in Intraocular Pressure
Description: Baseline and change from baseline at 6 months in intraocular pressure as measured by applanation tonometry
Time Frame: Baseline and 6 months
Population: The Intent-to-treat population included all subjects who received study treatment. No values were imputed for missing data.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | TX Naïve Arm | Previous TX Arm
Number analyzed (Participants) | 10 | 10
mm Hg
  Baseline | 14.2 (3.52) | 13.3 (2.50)
  Month 6: number analyzed (Participants) | 10 | 9
  Month 6 | -0.3 (2.41) | 2.8 (7.89)

3. Secondary Outcome: Mean Change From Baseline in Central Subfield Thickness
Description: Baseline and change from baseline at 6 months in central subfield thickness. Central subfield thickness (CST) is a diagnostic measurement used in identifying the presence of edema in the circular area 1 mm in diameter centered around the fovea. CST was measured using spectral domain optical coherence tomography (SD-OCT). A masked reading center graded the SD-OCT digital images. A negative change from baseline value represents a reduction in macular edema.
Time Frame: Baseline and 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Previous TX Arm | TX Naïve Arm
Number analyzed (Participants) | 10 | 10
Microns
  Baseline | 421.6 (94.33) | 472.7 (109.46)
  Month 6: number analyzed (Participants) | 10 | 9
  Month 6 | -90.9 (62.48) | -119.6 (65.48)

4. Secondary Outcome: Best Corrected Visual Acuity
Description: Baseline and Change from baseline at 6 months in best corrected visual acuity before and after treatment Best corrected visual acuity (BCVA) refers to the measurement of the best possible vision that can be achieved following refraction or correction. BCVA was assessed following the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol and was measured as the number of letters read correctly on an ETDRS eye chart. A positive change from baseline value represents an improvement in vision.
Time Frame: Baseline and 6 months
Population: The Intent-to-treat population included all subjects who received study treatment.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | TX Naïve Arm | Previous TX Arm
Number analyzed (Participants) | 10 | 10
Letters
  Baseline | 67.2 (11.66) | 67.2 (8.95)
  Month 6: number analyzed (Participants) | 10 | 9
  Month 6 | 8.5 (11.96) | 1.1 (11.94)

5. Secondary Outcome: CLS-TA Injections
Description: After the initial treatment with CLS-TA, with or without intravitreal aflibercept, at Baseline, retreatment with CLS-TA was allowed in either treatment group from Month 2 through Month 6 if pre-defined retreatment criteria were met. Number of patients receiving 0, 1, 2, 3, 4 or 5 retreatments with CLS-TA.
Time Frame: 2 to 6 months following initial treatment with study drug
Population: The Intent-to-treat population included all subjects who received study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | TX Naïve Arm | Previous TX Arm
Number analyzed (Participants) | 10 | 10
Participants
  0 additional injections | 4 | 1
  1 additional injection | 2 | 3
  2 additional injections | 0 | 2
  3 additional injections | 2 | 0
  4 additional injections | 2 | 4

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | TX Naïve Arm | Previous TX Arm
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 8/10 | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TX Naïve Arm (N=10) | Previous TX Arm (N=10)
Cataract (Eye disorders) | 3 (3) | 2 (2) — #Study eye
Cataract (Eye disorders) | 2 (2) | 0 (0) — #Fellow eye
Conjunctival haemorrhage (Eye disorders) | 3 (3) | 2 (2) — #Study eye
Dry eye (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Dry eye (Eye disorders) | 0 (0) | 1 (1) — #Fellow eye
Episcleritis (Eye disorders) | 0 (0) | 1 (1) — #Fellow eye
Eye irritation (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Eye irritation (Eye disorders) | 1 (1) | 0 (0) — #Fellow eye
Eye pain (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Iritis (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Macular fibrosis (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Ocular hypertension (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Intraocular pressure increased (Investigations) | 1 (1) | 0 (0) — #Study eye
Optic nerve cup/disc ratio increased (Investigations) | 0 (0) | 1 (1) — #Fellow eye
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The institution and investigators participating in this trial shall have no right to publish or present the results of this study without the prior written consent of Clearside Biomedical.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-23): https://cdn.clinicaltrials.gov/large-docs/24/NCT02949024/Prot_SAP_000.pdf